CLINICAL TRIAL: NCT06596603
Title: CAN-REST: Contrast-Associated Nephropathy Risk Evaluation in Acute Ischemic Stroke After Endovascular Thrombectomy
Brief Title: Contrast-Associated Nephropathy Risk Evaluation in Acute Ischemic Stroke After Endovascular Thrombectomy
Acronym: CAN-REST
Status: Completed | Type: Observational
Sponsor: Niguarda Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 4658_17.04.2024_N
Record Dates: First submitted 2024-08-28; First posted 2024-09-19 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Contrast-Associated Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The CAN-REST study is a multicenter, observational, and retrospective study aimed at evaluating the incidence and risk factors of contrast-associated acute kidney injury (CA-AKI) in patients with acute ischemic stroke (AIS) who undergo endovascular thrombectomy (EVT). This study is conducted across multiple centers in Italy, Europe, the USA, and Canada, and includes data from AIS patients treated with EVT in 2023. The primary objectives are to assess the incidence of CA-AKI in this population and identify associated risk factors. Secondary objectives include evaluating the impact of CA-AKI on clinical outcomes, such as the length of hospital stay, functional recovery, and 90-day mortality, as well as developing risk stratification tools to predict CA-AKI. By analyzing a large cohort of patients, CAN-REST aims to provide critical insights into the renal complications associated with EVT and establish predictive models that can guide clinical decision-making and improve patient outcomes.

DETAILED DESCRIPTION:
The CAN-REST study is a multicenter, observational, and retrospective study designed to evaluate the incidence and risk factors of contrast-associated acute kidney injury (CA-AKI) in patients who have suffered an acute ischemic stroke (AIS) and subsequently underwent endovascular thrombectomy (EVT). The use of contrast agents during EVT, essential for visualizing blood vessels and guiding the procedure, poses a risk for CA-AKI, particularly in patients who are already in a vulnerable state due to stroke-related comorbidities and the acute nature of their condition.

The primary objective of the study is to assess the incidence of CA-AKI in AIS patients following EVT and to identify specific risk factors that contribute to the development of CA-AKI. Secondary objectives include evaluating the impact of CA-AKI on clinical outcomes, such as the length of hospital stay, functional recovery as measured by the modified Rankin Scale (mRS) at discharge and 90 days post-procedure, and all-cause mortality at 90 days. Additionally, the study aims to develop and validate risk stratification tools that can predict the likelihood of CA-AKI based on both baseline patient characteristics and procedural variables related to EVT.

The study population consists of all consecutive AIS patients treated with EVT in participating centers from January 1, 2023, to December 31, 2023. Data collection will include detailed information on patient demographics, clinical history, stroke severity, procedural details of EVT, and subsequent renal function assessments to determine the development of CA-AKI. Two predictive models will be developed: one using only pre-EVT variables and another incorporating EVT-related variables to better stratify patients according to their risk for developing CA-AKI.

By analyzing a large cohort of patients from multiple centers worldwide, CAN-REST aims to provide valuable insights into the renal complications associated with the use of contrast media in EVT for AIS patients. The study's findings are expected to guide clinical practice by identifying high-risk patients and enabling the development of preventative strategies, ultimately improving patient outcomes and care standards in stroke treatment.

ELIGIBILITY:
To be eligible to participate in this study, subjects must meet all of the following criteria:

* Age >18 years at the time of AIS
* Documented serum creatinine:

  * pre-EVT and
  * within 48h and/or within 7 days after EVT. Patients on chronic dialysis will be collected but excluded from the analyses

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive EVT-treated acute ischemic stroke patients discharged at the participating centers from 1 January 2023 to 31 December 2023.
Sampling Method: Non-Probability Sample
Enrollment: 8000 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-07-01 (Actual)

PRIMARY OUTCOMES:
Incidence of Contrast-Associated Acute Kidney Injury (CA-AKI) | Within 48 hours and up to 7 days post-endovascular thrombectomy.
  Measure the occurrence of acute kidney injury characterized by an increase in serum creatinine ≥0.3 mg/dL or ≥50% within 48 hours, or an increase of ≥0.3 mg/dL within 7 days post-endovascular thrombectomy in acute ischemic stroke patients.

SECONDARY OUTCOMES:
Days of In-Hospital Stay | Measured daily from hospital admission until the day of discharge post-endovascular thrombectomy, assessed up to 30 days
  Measure the total number of days patients remain hospitalized following endovascular thrombectomy
Functional Recovery (modified Rankin Scale, mRS; ranging from 0 [full recovery] to 6[death]) | 90 days post-procedure
  Assess the level of disability or dependence in daily activities of patients post-stroke, measured at discharge and at 90 days post-procedure
All-Cause Mortality at 90 Days (modified Rankin Scale, mRS = 6) | 90 days post-procedure
  Measure the number of deaths from any cause within 90 days following endovascular thrombectomy Time Frame: 90 days post-procedure.
Development of Risk Stratification Tools | 24 hours, 48 hours, at 3 months, and at 12 months post-endovascular thrombectomy
  Create and validate predictive models for CA-AKI using baseline and EVT-related variables to categorize patients into risk groups (low, medium, high)

CONTACTS AND LOCATIONS:
Locations (1):
- ASST Grande Ospedale Metropolitano Niguarda, Milan, Lombardy, Italy

IPD SHARING:
Plan to Share IPD: No